CLINICAL TRIAL: NCT04644276
Title: Feasibility Study of a Mask Adhesive in Patients Treated With NIV in an Institutional Setting
Brief Title: Mask Adhesive Institutional Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Challenges with recruitment
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SRCHRCMask Adhesive 2020_11130
Record Dates: First submitted 2020-11-18; First posted 2020-11-25 (Actual); Results first posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Respiratory Failure; Covid19
MeSH Terms: conditions — Respiratory Insufficiency; COVID-19 | interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Mask with Mask Adhesive/Arm 1 (Active Comparator): Patients will be randomized to AF531 if they receive mask adhesive with mask on the first study night then the mask without mask adhesive(Performatrak) on the second study night.
  Interventions: Device: Mask with Mask Adhesive/Arm 1
- Mask without Mask Adhesive/Arm 2 (Placebo Comparator): Patients will be randomized to Arm 2 if they receive the mask without mask adhesive on the first study night then they will receive the mask with the mask adhesive on the second study night.
  Interventions: Device: Mask without Mask Adhesive / Arm 2

INTERVENTIONS:
Device: Mask with Mask Adhesive/Arm 1 — Patients will be randomized to Arm1 if they receive the mask adhesive and mask on the first study night then the mask without the mask adhesive on the second study night.
  Arms: Mask with Mask Adhesive/Arm 1
Device: Mask without Mask Adhesive / Arm 2 — Patients will be randomized to Arm 2 if they receive the mask without mask adhesive on the first study night then the mask adhesive with the mask on the second study night.
  Arms: Mask without Mask Adhesive/Arm 2

SUMMARY:
To reduce interface leak and aerosol spread, Philips has developed an accessory to non-invasive ventilation(NIV) masks to be used with the Philips AF531 and the PerformaTrak mask on respiratory failure patients. For the purposes of capturing initial mask leak and safety data, this trial will enroll patients treated with NIV in an institutional setting (i.e., sleep lab).

DETAILED DESCRIPTION:
The Mask Adhesive will serve as an accessory to the AF531/PerformaTrak masks with the intention to reduce patient leak while a patient is receiving therapy. This accessory is a double-sided adhesive; with one side applied directly to the patient's skin and the other side connected to the mask cushion. Each adhesive is only to be applied to a patient once. The AF531/Performatrak mask can be removed from the adhesive and then re-applied, as necessary. For example, if the patient needs to remove the mask to eat or take medicine, the mask is removed from the patient and the adhesive will stay on the patient's face

ELIGIBILITY:
Inclusion Criteria:

* Adults patients age 18 to 85 (inclusive)
* Adult patients treated with NIV
* Able to read, write, and speak English
* Able to provide written informed consent
* Willing to have facial hair removed for adhesive placement (if required)

Exclusion Criteria:

* Pre-existing allergy to tape or adhesive;
* Blisters, open skin or pre-existing skin condition that may impact the ability to support removal of the mask adhesive without tearing the skin
* pregnant (for females of childbearing age);
* Individuals sentenced to such an institution under a criminal or civil statute,
* Individuals detained in other facilities by virtue of statutes or commitment procedures which provide alternatives to criminal prosecution or incarceration in a penal institution, and individuals detained pending arraignment, trial, or sentencing

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Disorder Center of Alabama, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mask With Mask Adhesive Then Mask Without Mask Adhesive: Adult patients treated with NIV (Non-Invasive Ventilation). In Arm 1, patients were randomized to receive the mask with mask adhesive (Performatrak) on the first study night then the mask without mask adhesive on the second study night. Due to the small sample size baseline data was not broken out by randomized order.
- Mask Without Mask Adhesive Then Mask With Mask Adhesive: Adult patients treated with NIV (Non-Invasive Ventilation). In Arm 2, patients were randomized to receive the mask without mask adhesive on the first study night then the mask with mask adhesive (Performatrak) on the second study night. Due to the small sample size baseline data was not broken out by randomized order.
- Clinician Participants: Clinicians will apply the mask adhesive to the participants and will complete ease-of-use measures.
Period: Overall Study
Arm/Group | Mask With Mask Adhesive Then Mask Without Mask Adhesive | Mask Without Mask Adhesive Then Mask With Mask Adhesive | Clinician Participants
Started | 2 | 3 | 2
Completed | 2 | 3 | 1
Not Completed | 0 | 0 | 1
Not completed — Did not complete overall impressions as study was put on hold and then terminated | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Adult patients treated with NIV (Non-Invasive Ventilation). Patients wore the AF541 mask with or without mask adhesive for one night in randomized order. Since this was a crossover study with so few participants, baseline data was presented for the overall patient population. Demographic data was not collected for clinician participants, so baseline data is not available.
Groups:
- Patient Participants: Adult patients treated with NIV (Non-Invasive Ventilation)
Arm/Group | Patient Participants
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Medical Adhesive-Related Skin Injury (MARSI)
Description: Percentage of patients who have severe and extreme skin irritation that persists for ≥ 30 min after mask adhesive removal (score of ≥ 3 on a 5-point grading system).
Time Frame: Up to 5 business days
Measure: Count of Participants; unit: Participants
Groups:
- Mask With Mask Adhesive: Results for Mask with Mask Adhesive intervention
- Mask Without Mask Adhesive: Results for Mask without Mask Adhesive intervention
Arm/Group | Mask With Mask Adhesive | Mask Without Mask Adhesive
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

2. Primary Outcome: Clinician Ease of Use
Description: Clinician-perceived mask adhesive ease-of-use as measured by a 0-10 Likert Scale at baseline (initial impressions) and study completion (overall impressions) Specifically, the item, "How would you rate the ease of application of the adhesive to the mask?" (On a 0 to 10 scale, with 0=Extremely Difficult and 10=Extremely Easy)
Time Frame: Initial Impressions at Baseline and Overall Impressions at Study Completion (After at least two mask applications)
Population: One participant did not complete overall impressions due to study on hold and then terminated.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinician Participants
Number analyzed (Participants) | 2
units on a scale
  Initial Impressions | 10 (0)
  Overall Impressions: number analyzed (Participants) | 1
  Overall Impressions | 10 (NA) — N=1

3. Secondary Outcome: Leak Change
Description: Change in leak volume (L/min) after mask adhesive use as compared to the use of the mask without the adhesive. Percent change in leak (endpoint per protocol) is reported in the Statistical Analysis section.
Time Frame: Up to 5 business days
Population: Absolute within-subject difference in leak: [Mask with mask adhesive] - [Mask without mask adhesive]
Measure: Median (Full Range); unit: Liters per minute
Groups:
- Mask With Mask Adhesive: Results for the Mask with Mask Adhesive intervention.
- Mask Without Mask Adhesive: Results for the Mask without Mask Adhesive intervention.
- Absolute Within-Subject Difference in Leak: Absolute Within-Subject Difference in Leak: [Leak from Mask with mask adhesive] - [Leak from Mask without mask adhesive]
Arm/Group | Mask With Mask Adhesive | Mask Without Mask Adhesive | Absolute Within-Subject Difference in Leak
Number analyzed (Participants) | 5 | 5 | 5
Liters per minute | 3.3 [0.2 to 19.9] | 3.2 [0.4 to 49.6] | -0.1 [-29.7 to 4.5]
Statistical Analysis 1: Comparison: Mask With Mask Adhesive vs Mask Without Mask Adhesive; Percent change in leak 100% x ([Mask with mask adhesive] - [Mask without mask adhesive])/ [Mask without mask adhesive]. The comparison between the two arms is captured in the reported percentage change; Test type: Superiority; p = 0.8125, Wilcoxon Signed-Ranks test; Median Difference (Final Values) = -37, 95% CI 2-sided [-112.6 to 140.7], Standard Deviation 102 — Unit is percent change

ADVERSE EVENTS:
Time Frame: Duration of study participation (Up to five business days from beginning to end of study)
Groups:
- Patient Participants: Adult patients treated with NIV (Non-Invasive Ventilation) No adverse events were reported, therefore, there was no need to compare the frequency of AEs between treatment arms. Adverse events were not collected for Clinicians participants.
Arm/Group | Patient Participants
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/76/NCT04644276/Prot_SAP_000.pdf